CLINICAL TRIAL: NCT00686595
Title: swiTching From etAnercept to iNfliximab in the Treatment of Moderate to Severe Psoriasis; a Multi-center, Open Label Trial evaluatinG the Efficacy, tOlerance and Safety (TANGO)
Brief Title: A Study to Evaluate the Switch From Etanercept to Infliximab in Subjects With Moderate-to-Severe Psoriasis (Study P05133)
Acronym: TANGO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Centocor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P05133; 2007-000535-26 (EudraCT Number)
Record Dates: First submitted 2008-05-27; First posted 2008-05-30 (Estimated); Results first posted 2011-02-24 (Estimated); Last update posted 2023-08-09 (Actual); Status verified 2023-07

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Infliximab 5 mg/kg (Experimental): Infliximab 5 mg/kg intravenous (IV) infusion administered at Baseline (Week 0), Visit 3 (Week 2), Visit 4 (Week 6), Visit 6 (Week 14), and Visit 8 (Week 22).
  Interventions: Biological: Infliximab

INTERVENTIONS:
Biological: Infliximab — Infliximab 5 mg/kg IV infusion.
  Other Names: Remicade, SCH 215596

SUMMARY:
This study will evaluate the efficacy, tolerability, and effect on the quality of life of infliximab in adults with moderate-to-severe psoriasis who are resistant to etanercept after 12 weeks of treatment or have failed 24 weeks of treatment with etanercept. Infliximab will be administered as an intravenous infusion of 5 mg/kg at Baseline (Week 0), Visit 3 (Week 2), Visit 4 (Week 6), Visit 6 (Week 14), and Visit 8 (Week 22).

ELIGIBILITY:
Inclusion Criteria:

* >=18 to 75 years of age at Screening, either sex, and any race.
* Diagnosis of moderate-to-severe plaque psoriasis >6 months prior to Screening.
* Resistant (after 12 weeks) or failed 24 weeks of etanercept treatment.
* Not reached PASI 75 at Screening Visit after 24 weeks of etanercept treatment or resistant to etanercept.
* Agree to avoid prolonged sun exposure or artificial ultraviolet light sources during study.
* Satisfy requirements of Screening and tuberculosis (TB) test as specified in protocol.
* Chest x-ray at Visit 1 or within 3 months prior to Visit 1 with no evidence of malignancy, infection, or fibrosis.
* Laboratory tests must be within protocol-specified parameters.
* Free of any clinically significant disease that would interfere with study evaluations.
* Willing to participate and adhere to study procedures by signing written informed consent.
* Women of childbearing potential and all men must be using adequate birth control measures and continue to do so until 6 months after receiving last dose of study medication.
* Females of childbearing potential must have negative serum pregnancy test at Visit 1 and negative urine pregnancy test at Visit 2.

Exclusion Criteria:

* Achieve PASI 75 or have BSA <10% after 24 weeks of etanercept.
* Current drug-induced psoriasis.
* Females who are pregnant or nursing and both males and females who are planning pregnancy during study period or during 6 months after receiving last dose of study medication.
* Previously treated with infliximab.
* Currently taking or have taken protocol-specified prohibited drugs within specified time frame prior to Baseline.
* Congestive Heart Failure (CHF)
* Chronic or recurrent infectious disease.
* Have or have had serious infection, or been hospitalized or received IV antibiotics for this infection during the 2 months prior to Visit 1.
* Have or have had opportunistic infection within 6 months prior to Visit 1.
* Have or have had herpes zoster infection within 2 months prior to Visit 1.
* Human Immunodeficiency Virus (HIV), hepatitis B or C.
* History of any clinically significant adverse events (AEs) to murine or chimeric proteins or human/murine recombinant products.
* Current signs or symptoms of severe, progressive, or uncontrolled renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, cardiac, neurological, cerebral, or psychiatric disease.
* History of demyelinating disease or symptoms suggestive of multiple sclerosis or optic neuritis.
* Current signs and symptoms or history of systemic lupus erythematosus.
* Transplanted organ (exception - corneal transplant >3 months prior to Visit 1).
* History of lymphoproliferative disease, including lymphoma, or signs and symptoms suggestive of possible lymphoproliferative disease, such as lymphadenopathy of unusual size or location.
* Malignancy within previous 5 years (exception - basal cell carcinoma of skin that has been treated with no evidence of recurrence).
* Unable or unwilling to undergo multiple venipunctures because of poor tolerability or lack of easy access to veins.
* Have had substance abuse (drug or alcohol) problem within previous 3 years.
* History of any clinically significant adverse reactions (including allergic reactions) to paracetamol/acetaminophen or histamine H1 receptor antagonist.
* In a situation or have a condition that, in opinion of investigator, may interfere with optimal participation in study.
* Used investigational drugs within 4 weeks of Screening.
* Participating in any other clinical study.
* Staff personnel directly involved with this study.
* Family members of investigational study staff.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2007-10-01 (Actual); Primary Completion 2009-10-01 (Actual); Study Completion 2009-10-01 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Ayala F, Lambert J; TANGO Study Group. Efficacy, tolerability and safety of switching from etanercept to infliximab for the treatment of moderate-to-severe psoriasis: A multicenter, open-label trial (TANGO). J Dermatolog Treat. 2015;26(4):304-11. doi: 10.3109/09546634.2014.952611. Epub 2014 Sep 18. PMID 25231176

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 48 participants were enrolled in this study. Of these, 38 participants received at least one dose of the study medication and represent the intent-to-treat (ITT) population.
Groups:
- Infliximab 5 mg/kg: Infliximab 5 mg/kg IV administered at Baseline (Week 0), Visit 3 (Week 2), Visit 4 (Week 6), Visit 6 (Week 14), and Visit 8 (Week 22).
Period: Overall Study
Arm/Group | Infliximab 5 mg/kg
Started | 38
Completed | 31
Not Completed | 7
Not completed — Adverse Event | 3
Not completed — Protocol Violation | 1
Not completed — Lost to Follow-up | 1
Not completed — Lack of Efficacy | 1
Not completed — Poor Compliance | 1

BASELINE CHARACTERISTICS:
Arm/Group | Infliximab 5 mg/kg
Number analyzed (Participants) | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.54 (9.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 28

OUTCOME MEASURES:

1. Primary Outcome: Psoriasis Area and Severity Index (PASI) 75 Response Rate at Week 10
Description: PASI correlates to the physician's assessment of psoriasis symptoms including redness of lesions, thickness of lesions, scaliness of lesions and extent of disease. Each parameter is graded from 0-4, 0 refers to no disease and 4 to severe involvement. The body is divided into 4 areas for scoring (head, arms, trunk to groin, legs to top of buttocks), and the final score ranges from 0-72. The PASI 75 response rate at Week 10 is measured as the percentage of participants who achieved at least 75% improvement from baseline PASI at Week 10.
Time Frame: Baseline and 10 weeks
Population: Participants from the intent-to-treat (ITT) population for whom the PASI assessment was available.
Measure: Number; unit: Percentage of participants
Arm/Group | Infliximab 5 mg/kg
Number analyzed (Participants) | 35
Percentage of participants | 71

2. Secondary Outcome: PASI 75 Response Rate at Week 18
Description: PASI correlates to the physician's assessment of psoriasis symptoms including redness of lesions, thickness of lesions, scaliness of lesions and extent of disease. Each parameter is graded from 0-4, 0 refers to no disease and 4 to severe involvement. The body is divided into 4 areas for scoring (head, arms, trunk to groin, legs to top of buttocks), and the final score ranges from 0-72. The PASI 75 response rate at Week 18 is measured as the percentage of participants who achieved at least 75% improvement from baseline PASI at Week 18.
Time Frame: Baseline and 18 weeks
Population: Participants from the ITT population for whom the PASI assessment was available.
Measure: Number; unit: Percent of participants
Arm/Group | Infliximab 5 mg/kg
Number analyzed (Participants) | 32
Percent of participants | 94

3. Secondary Outcome: PASI 75 Response Rate at Week 24
Description: PASI correlates to the physician's assessment of psoriasis symptoms including redness of lesions, thickness of lesions, scaliness of lesions and extent of disease. Each parameter is graded from 0-4, 0 refers to no disease and 4 to severe involvement. The body is divided into 4 areas for scoring (head, arms, trunk to groin, legs to top of buttocks), and the final score ranges from 0-72. The PASI 75 response rate at Week 24 is measured as the percentage of participants who achieved at least 75% improvement from baseline PASI at Week 24.
Time Frame: Baseline and 24 weeks
Population: Participants from the ITT population for whom the PASI assessment was available.
Measure: Number; unit: Percentage of participants
Arm/Group | Infliximab 5 mg/kg
Number analyzed (Participants) | 35
Percentage of participants | 74

4. Secondary Outcome: PASI 50 Response Rate at Week 10
Description: PASI correlates to the physician's assessment of psoriasis symptoms including redness of lesions, thickness of lesions, scaliness of lesions and extent of disease. Each parameter is graded from 0-4, 0 refers to no disease and 4 to severe involvement. The body is divided into 4 areas for scoring (head, arms, trunk to groin, legs to top of buttocks), and the final score ranges from 0-72. The PASI 50 response rate at Week 10 is measured as the percentage of participants who achieved at least 50% improvement from baseline PASI at Week 10.
Time Frame: Baseline and 10 weeks
Population: Participants from the ITT population for whom the PASI assessment was available.
Measure: Number; unit: Percentage of participants
Arm/Group | Infliximab 5 mg/kg
Number analyzed (Participants) | 35
Percentage of participants | 91

5. Secondary Outcome: PASI 50 Response Rate at Week 18
Description: PASI correlates to the physician's assessment of psoriasis symptoms including redness of lesions, thickness of lesions, scaliness of lesions and extent of disease. Each parameter is graded from 0-4, 0 refers to no disease and 4 to severe involvement. The body is divided into 4 areas for scoring (head, arms, trunk to groin, legs to top of buttocks), and the final score ranges from 0-72. The PASI 50 response rate at Week 18 is measured as the percentage of participants who achieved at least 50% improvement from baseline PASI at Week 18.
Time Frame: Baseline and 18 weeks
Population: Participants from the ITT population for whom the PASI assessment was available.
Measure: Number; unit: Percentage of participants
Arm/Group | Infliximab 5 mg/kg
Number analyzed (Participants) | 32
Percentage of participants | 97

6. Secondary Outcome: PASI 50 Response Rate at Week 24
Description: PASI correlates to the physician's assessment of psoriasis symptoms including redness of lesions, thickness of lesions, scaliness of lesions and extent of disease. Each parameter is graded from 0-4, 0 refers to no disease and 4 to severe involvement. The body is divided into 4 areas for scoring (head, arms, trunk to groin, legs to top of buttocks), and the final score ranges from 0-72. The PASI 50 response rate at Week 24 is measured as the percentage of participants who achieved at least 50% improvement from baseline PASI at Week 24.
Time Frame: Baseline and 24 weeks
Population: Participants from the ITT population for whom the PASI assessment was available.
Measure: Number; unit: Percentage of participants
Arm/Group | Infliximab 5 mg/kg
Number analyzed (Participants) | 35
Percentage of participants | 89

7. Secondary Outcome: PASI 90 Response Rate at Week 10
Description: PASI correlates to the physician's assessment of psoriasis symptoms including redness of lesions, thickness of lesions, scaliness of lesions and extent of disease. Each parameter is graded from 0-4, 0 refers to no disease and 4 to severe involvement. The body is divided into 4 areas for scoring (head, arms, trunk to groin, legs to top of buttocks), and the final score ranges from 0-72. The PASI 90 response rate at Week 10 is measured as the percentage of participants who achieved at least 90% improvement from baseline PASI at Week 10.
Time Frame: Baseline and 10 weeks
Population: Participants from the ITT population for whom the PASI assessment was available.
Measure: Number; unit: Percentage of participants
Arm/Group | Infliximab 5 mg/kg
Number analyzed (Participants) | 35
Percentage of participants | 37

8. Secondary Outcome: PASI 90 Response Rate at Week 18
Description: PASI correlates to the physician's assessment of psoriasis symptoms including redness of lesions, thickness of lesions, scaliness of lesions and extent of disease. Each parameter is graded from 0-4, 0 refers to no disease and 4 to severe involvement. The body is divided into 4 areas for scoring (head, arms, trunk to groin, legs to top of buttocks), and the final score ranges from 0-72. The PASI 90 response rate at Week 18 is measured as the percentage of participants who achieved at least 90% improvement from baseline PASI at Week 18.
Time Frame: Baseline and 18 weeks
Population: Participants from the ITT population for whom the PASI assessment was available.
Measure: Number; unit: Percentage of participants
Arm/Group | Infliximab 5 mg/kg
Number analyzed (Participants) | 32
Percentage of participants | 56

9. Secondary Outcome: PASI 90 Response Rate at Week 24
Description: PASI correlates to the physician's assessment of psoriasis symptoms including redness of lesions, thickness of lesions, scaliness of lesions and extent of disease. Each parameter is graded from 0-4, 0 refers to no disease and 4 to severe involvement. The body is divided into 4 areas for scoring (head, arms, trunk to groin, legs to top of buttocks), and the final score ranges from 0-72. The PASI 90 response rate at Week 24 is measured as the percentage of participants who achieved at least 90% improvement from baseline PASI at Week 24.in PASI at Week 24
Time Frame: Baseline and 24 weeks
Population: Participants from the ITT population for whom the PASI assessment was available.
Measure: Number; unit: Percentage of participants
Arm/Group | Infliximab 5 mg/kg
Number analyzed (Participants) | 35
Percentage of participants | 54

10. Secondary Outcome: PASI 100 Response Rate at Week 10
Description: PASI correlates to the physician's assessment of psoriasis symptoms including redness of lesions, thickness of lesions, scaliness of lesions and extent of disease. Each parameter is graded from 0-4, 0 refers to no disease and 4 to severe involvement. The body is divided into 4 areas for scoring (head, arms, trunk to groin, legs to top of buttocks), and the final score ranges from 0-72. The PASI 100 response rate at Week 10 is measured as the percentage of participants who achieved 100% improvement from baseline PASI at Week 10.
Time Frame: Baseline and 10 weeks
Population: Participants from the ITT population for whom the PASI assessment was available.
Measure: Number; unit: Percentage of participants
Arm/Group | Infliximab 5 mg/kg
Number analyzed (Participants) | 35
Percentage of participants | 17

11. Secondary Outcome: PASI 100 Response Rate at Week 18
Description: PASI correlates to the physician's assessment of psoriasis symptoms including redness of lesions, thickness of lesions, scaliness of lesions and extent of disease. Each parameter is graded from 0-4, 0 refers to no disease and 4 to severe involvement. The body is divided into 4 areas for scoring (head, arms, trunk to groin, legs to top of buttocks), and the final score ranges from 0-72. The PASI 100 response rate at Week 18 is measured as the percentage of participants who achieved 100% improvement from baseline PASI at Week 18.
Time Frame: Baseline and 18 weeks
Population: Participants from the ITT population for whom the PASI assessment was available.
Measure: Number; unit: Percentage of participants
Arm/Group | Infliximab 5 mg/kg
Number analyzed (Participants) | 32
Percentage of participants | 31

12. Secondary Outcome: PASI 100 Response Rate at Week 24
Description: PASI correlates to the physician's assessment of psoriasis symptoms including redness of lesions, thickness of lesions, scaliness of lesions and extent of disease. Each parameter is graded from 0-4, 0 refers to no disease and 4 to severe involvement. The body is divided into 4 areas for scoring (head, arms, trunk to groin, legs to top of buttocks), and the final score ranges from 0-72. The PASI 100 response rate at Week 24 is measured as the percentage of participants who achieved 100% improvement from baseline PASI at Week 24.
Time Frame: 24 weeks
Population: Participants from the ITT population for whom the PASI assessment was available.
Measure: Number; unit: Percentage of participants
Arm/Group | Infliximab 5 mg/kg
Number analyzed (Participants) | 35
Percentage of participants | 40

13. Secondary Outcome: Percent Reduction in Self-Administered Psoriasis Area Severity Index (SAPASI) at Week 18
Description: SAPASI is the participant's measurement of severity of psoriasis. The participant estimates the area of psoriatic involvement for each body district (head, upper limbs, trunk and lower limbs) and scores it from 0 (no involvement)-6 (90-100% involvement); and the extent of psoriasis from 0 (no involvement) to 4 (very marked) for each - erythema, desquamation and induration of the plaques. The final score computed by the investigator ranged from 0-72. The percent reduction in SAPASI at Week 18 compared to baseline is reported.
Time Frame: Baseline and Week 18
Population: Participants from the ITT population for whom the SAPASI assessment was available.
Measure: Mean (Standard Deviation); unit: Percent reduction
Arm/Group | Infliximab 5 mg/kg
Number analyzed (Participants) | 31
Percent reduction | 89 (15)

14. Secondary Outcome: Percent Reduction in SAPASI at Week 24
Description: SAPASI is the participant's measurement of severity of psoriasis. The participant estimates the area of psoriatic involvement for each body district (head, upper limbs, trunk and lower limbs) and scores it from 0 (no involvement)-6 (90-100% involvement); and the extent of psoriasis from 0 (no involvement) to 4 (very marked) for each - erythema, desquamation and induration of the plaques. The final score computed by the investigator ranged from 0-72. The percent reduction in SAPASI at Week 24 compared to baseline is reported.
Time Frame: Baseline and Week 24
Population: Participants from the ITT population for whom the SAPASI assessment was available.
Measure: Mean (Standard Deviation); unit: Percent reduction
Arm/Group | Infliximab 5 mg/kg
Number analyzed (Participants) | 33
Percent reduction | 82 (29)

15. Secondary Outcome: Percent Reduction in Affected Body Surface Area (BSA) at Week 18
Description: The BSA is the physician's evaluation for the extent of disease. The entire body area is divided into 4 districts: head, upper limbs, trunk and lower limbs to which corresponds the 10%, 20%, 30% and 40% of the entire body surface respectively. The investigator assesses the percentage of the participant's body surface area affected by psoriasis in each district. The final affected BSA value is the sum of the percentage of each district. The percent reduction in affected BSA at Week 18 compared to baseline is reported.
Time Frame: Baseline and Week 18
Population: Participants from the ITT population for whom the BSA assessment was available.
Measure: Mean (Standard Deviation); unit: Percent reduction
Arm/Group | Infliximab 5 mg/kg
Number analyzed (Participants) | 32
Percent reduction | 82 (28)

16. Secondary Outcome: Percent Reduction in Affected BSA at Week 24
Description: The BSA is the physician's evaluation for the extent of disease. The entire body area is divided into 4 districts: head, upper limbs, trunk and lower limbs to which corresponds the 10%, 20%, 30% and 40% of the entire body surface respectively. The investigator assesses the percentage of the participant's body surface area affected by psoriasis in each district. The final affected BSA value is the sum of the percentage of each district. The percent reduction in affected BSA at Week 24 compared to baseline is reported.
Time Frame: Baseline and Week 24
Population: Participants from the ITT population for whom the BSA assessment was available.
Measure: Mean (Standard Deviation); unit: Percent reduction
Arm/Group | Infliximab 5 mg/kg
Number analyzed (Participants) | 35
Percent reduction | 72 (39)

17. Secondary Outcome: Percent Reduction in Visual Analogue Scale (VAS) Referred Itch at Week 18
Description: VAS was used to measure itch. Participants reported itch using VAS - a line ranging from 0 cm to 10 cm, measured by the investigator. 0 cm referred to absence of itch and 10 cm referred to severe itching. The percent reduction in VAS at Week 18 compared to baseline is reported.
Time Frame: Baseline and Week 18
Population: Participants from the ITT population for whom the VAS assessment was available.
Measure: Mean (Standard Deviation); unit: Percent reduction
Arm/Group | Infliximab 5 mg/kg
Number analyzed (Participants) | 30
Percent reduction | 81 (27)

18. Secondary Outcome: Percent Reduction in VAS Referred Itch at Week 24
Description: VAS was used to measure itch. Participants reported itch using VAS - a line ranging from 0 cm to 10 cm, measured by the investigator. 0 cm referred to absence of itch and 10 cm referred to severe itching. The percent reduction in VAS at Week 24 compared to baseline is reported.
Time Frame: Baseline and Week 24
Population: Participants from the ITT population for whom the VAS assessment was available.
Measure: Mean (Standard Deviation); unit: Percent reduction
Arm/Group | Infliximab 5 mg/kg
Number analyzed (Participants) | 33
Percent reduction | 72 (38)

19. Secondary Outcome: Percent Reduction in Dermatology Life Quality Index (DLQI) Total Score at Week 18
Description: DLQI total score comprises 6 different aspects that may affect quality of life: symptoms and feelings, daily activities, leisure, work or school performance, personal relationships, and treatment. DLQI total scores range from 0 to 30, with 0 corresponding to the best quality of life and 30 to the worst. The percent reduction in DLQI score at Week 18 compared to baseline is reported.
Time Frame: Baseline and Week 18
Population: Participants from the ITT population for whom the DLQI assessment was available.
Measure: Mean (Standard Deviation); unit: Percent reduction
Arm/Group | Infliximab 5 mg/kg
Number analyzed (Participants) | 30
Percent reduction | 77 (35)

20. Secondary Outcome: Percent Reduction in DLQI Total Score at Week 24
Description: DLQI total score comprises 6 different aspects that may affect quality of life: symptoms and feelings, daily activities, leisure, work or school performance, personal relationships, and treatment. DLQI total scores range from 0 to 30, with 0 corresponding to the best quality of life and 30 to the worst. The percent reduction in DLQI score at Week 24 compared to baseline is reported.
Time Frame: Baseline and Week 24
Population: Participants from the ITT population for whom the DLQI assessment was available.
Measure: Mean (Standard Deviation); unit: Percent reduction
Arm/Group | Infliximab 5 mg/kg
Number analyzed (Participants) | 31
Percent reduction | 68 (50)

21. Secondary Outcome: Percent Reduction in Skin Index Questionnaire (SKINDEX-29) Score at Week 18
Description: The SKINDEX-29 measures the quality of life in dermatological participants, who complete a questionnaire assessing 3 scales - burden of symptoms, social functioning and emotional state. Participants answered 29 questions referring to the previous 4-week period, on a 5-point scale from "never" (=0) to "all the time" (=4). The score for each scale ranges from 0 to 100 and higher scores reflect a worse quality of life. The percent reduction in SKINDEX-29 scores at Week 18 compared to baseline is reported.
Time Frame: Baseline and Week 18
Population: Participants from the ITT population for whom the SKINDEX-29 assessments were available.
Measure: Mean (Standard Deviation); unit: Percent reduction
Arm/Group | Infliximab 5 mg/kg
Number analyzed (Participants) | 31
Percent reduction
  Symptoms score | 42 (26)
  Emotional state score | 39 (25)
  Social functioning score | 39 (27)

22. Secondary Outcome: Percent Reduction in SKINDEX-29 Scores at Week 24
Description: The SKINDEX-29 measures the quality of life in dermatological participants, who complete a questionnaire assessing 3 scales - burden of symptoms, social functioning and emotional state. Participants answered 29 questions referring to the previous 4-week period, on a 5-point scale from "never" (=0) to "all the time" (=4). The score for each scale ranges from 0 to 100 and higher scores reflect a worse quality of life. The percent reduction in SKINDEX-29 scores at Week 24 compared to baseline is reported.
Time Frame: Baseline and Week 24
Population: Participants from the ITT population for whom the SKINDEX-29 assessments were available.
Measure: Mean (Standard Deviation); unit: Percent reduction
Arm/Group | Infliximab 5 mg/kg
Number analyzed (Participants) | 34
Percent reduction
  Symptoms score | 40 (29)
  Emotional state score | 32 (34)
  Social functioning score | 31 (36)

ADVERSE EVENTS:
Arm/Group | Infliximab 5 mg/kg
Serious Adverse Events (participants affected / at risk) | 7/38
Other Adverse Events (participants affected / at risk) | 12/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infliximab 5 mg/kg (N=38)
Mitral Valve Prolapse (Cardiac disorders) | 1 (1)
Cyst (General disorders) | 1 (1)
Electrocution (General disorders) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 3 (4)
Completed Suicide (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infliximab 5 mg/kg (N=38)
Gastritis (Gastrointestinal disorders) | 2 (2)
Bronchitis (Infections and infestations) | 2 (2)
Rhinitis (Infections and infestations) | 3 (3)
Blood Triglycerides Increased (Investigations) | 2 (2)
Transaminases Increased (Investigations) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator agrees not to publish or publicly present any of the

study results without prior written authorization from sponsor, except than for the dispositions provided in the Minister's Decree and Ministerial Circular. Investigator agrees to provide 45 days written notice to sponsor prior to submission for publication or presentation to permit sponsor to review copies of abstracts/manuscripts for publication (including text for oral presentations) which report any study results.